CLINICAL TRIAL: NCT04865666
Title: Examining the Real-World Effectiveness of the Movr mHealth Application: A Mixed-Methods Pilot Pragmatic Randomized Controlled Trial
Brief Title: Examining the Real-World Effectiveness of the Movr App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Mitacs (Industry); Lululemon Athletica (Unknown)
Responsible Party: Principal Investigator, Mary Jung, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H19-01915
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Healthy
Keywords: mHealth; functional movement; flexibility; strength; cardiovascular fitness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- movr App Group (Experimental): Participants were instructed to maintain their usual physical activity, diet, and sleep behavior for the 8-week intervention period and to avoid any specialized exercise training for that time period, but they were also asked to use the movr app to supplement their current activity.
  Interventions: Device: movr mHealth App
- Waitlist Control Group (No Intervention): Participants were instructed to maintain their usual physical activity, diet, and sleep behavior over the 8-week study period and to avoid any specialized exercise training for that time period. Following the 8-week study period, individuals in the control group were permitted to download and use the movr app if they chose to.

INTERVENTIONS:
Device: movr mHealth App — The exercises prescribed through the movr app were accompanied with videos, images, and detailed instructions on how to complete them. These exercises consisted of basic movement and mobility patterns and are designed to promote functional movement. Participants were instructed to complete a total of four 'Minis' and two workout 'Builder' sessions per week. Workout Builders are designed to be longer exercise sessions tailored to the user's desired exercise time (15, 30, 45 or 60 min), equipment available (TRX Band, kettlebell, chin-up bar, dumbbells, foam roller, or none), target body region (lower, upper, or whole body), and specific exercise goal ('get sweaty,' 'build strength,' or 'develop mobility'). Version 3.6 of the movr app was used at the start of data collection and was updated to Version 4.1 over the course of the trial. No significant changes were made to the app or to the exercise prescription functionality throughout those updates.
  Arms: movr App Group

SUMMARY:
The objective of this 8-week pilot pragmatic randomized controlled trial was to examine the real-world impact of movr on functional movement, flexibility, strength, and cardiovascular fitness.

DETAILED DESCRIPTION:
Thousands of mobile apps available for download are geared towards health and fitness, yet limited research has evaluated the real-world effectiveness of such apps. The movr app is an mHealth app designed to enhance physical functioning by prescribing functional movement training based on individualized movement assessments. movr's influence on functional movement and physical fitness (flexibility, strength, and cardiovascular fitness) has not yet been established empirically. Thus, the objective of this 8-week pilot pragmatic randomized controlled trial was to examine the real-world impact of movr on functional movement, flexibility, strength, and cardiovascular fitness.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 50 years
* Ability to read and write English
* Owned a mobile device that could download applications from the App Store or Google Play

Exclusion Criteria:

* Previously used the movr app
* Had any contraindications to exercise based on the Get Active Questionnaire

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline in functional movement screen (FMS) at 8-week follow-up | Baseline and 8-week follow-up
  The 100-point version of the functional movement screen (FMS) was used to identify individual movement patterns. The FMS is a screening tool to assess full body movement patterns and consists of seven core movement tests (deep squat, hurdle step, in-line lunge, active straight-leg raise, shoulder flexibility, trunk stability push-up, and quadruped rotary stability). The seven FMS movement screens were performed by each participant and recorded using a portable observation lab (Noldus) with two video cameras (one shot on a sagittal plane [side] view and the other from a frontal plane [front/back] view). The standardized FMS verbal instructions were provided by the researcher. The video-based testing was completed to minimize participant burden during lab visits and to blind participants to their FMS scores for each of the movements. Scoring of the FMS was completed at a later time using the video recordings.

SECONDARY OUTCOMES:
Change from baseline in flexibility at 8-week follow-up | Baseline and 8-week follow-up
  The shoulder reach flexibility test was used to assess upper body flexibility and the sit and reach, active straight-leg raise (ASLR), and the half-kneeling dorsiflexion tests were used to assess lower body flexibility. For the shoulder reach test, a soft tape measure was used to measure the distance between participants' closed fists, and for the ASLR, range of motion in degrees were measured on each leg using a digital inclinometer (Metriks, Canada). For each of the flexibility tests (excluding sit and reach), scores from the left and right side (arm or leg) were summed and total scores are reported. A lower measurement score on the shoulder flexibility test indicates greater flexibility, while higher scores on the sit and reach, ASLR, and half-kneeling dorsiflexion tests indicate greater flexibility.
Change from baseline in muscular endurance at 8-week follow-up | Baseline and 8-week follow-up
  A push-up test was used to determine the maximal number of successive push-up repetitions that participants could complete until failure. The test protocols followed the Canadian Society for Exercise Physiology (CSEP) recommendations, including use of a modified push-up protocol for all women in the study.
Change from baseline in handgrip strength at 8-week follow-up | Baseline and 8-week follow-up
  Handgrip strength was assessed using a maximal voluntary contraction of an isometric handgrip squeeze using a Smedley spring handgrip dynamometer (BASELINE®). Scores from the left and right hand were summed and total scores are reported.
Change from baseline in lower body power at 8-week follow-up | Baseline and 8-week follow-up
  A countermovement jump (CMJ) was conducted using the My Jump 2 mobile app on an iPhone 8 to assess lower body power. The validity and reliability of the My Jump 2 has been established previously.
Change from baseline in cardiovascular fitness at 8-week follow-up | Baseline and 8-week follow-up
  Participants performed an incremental maximal oxygen uptake (V̇O2max) test on a cycle ergometer (Lode Excalibur Sport). The resistance on the cycle ergometer was automatically increased (1W every 3 s for women, 1W every 2 s for men) until participants reached volitional exhaustion or could no longer maintain a pedal cadence of at least 50 rpm. A metabolic cart with an online gas collection system (Parvo Medics, TrueOne 2400) was used to collect expired gas samples continuously and V̇O2max was calculated using the mean of the highest average oxygen consumption over a 30-s period (in mL·kg-1·min-1).
Changes from baseline in health locus of control at 8-week follow-up | Baseline and 8-week follow-up
  Form B of the Multidimensional Health Locus of Control Scale was used to measure health locus of control
Changes from baseline in perceptions of health at 8-week follow-up | Baseline and 8-week follow-up
  The Short Form (36) Health Survey was used to assess perceptions of health status
Changes from baseline in physical activity enjoyment at 8-week follow-up | Baseline and 8-week follow-up
  Enjoyment of physical activity completed over the past week was measured pre- and post-intervention using the Physical Activity Enjoyment Scale (PACES). This scale has 18 items that participants rated on a 7-point bipolar scale (from 1 to 7).
Changes from baseline in well-being, enjoyment, satisfaction with physical functioning at 1, 2, 3, 4, 5, 6, 7, and 8-week follow-up | Baseline and 1, 2, 3, 4, 5, 6, 7, and 8-week follow-up
  The Subjective Exercise Experiences Scale (SEES) was used to measure participants' positive well-being, psychological distress and fatigue. The single-item Exercise Enjoyment Scale (EES) was used to measure exercise enjoyment. A 5-item measure of satisfaction with physical functioning was used assess participants' satisfaction with their (1) overall physical functioning, (2) cardiovascular fitness, (3) muscle strength, (4) flexibility, and (5) balance. This set of questions was administered at the end of each week throughout the 8-week intervention period as well as pre- and post-intervention in the form of an email that included a Qualtrics link to the survey
Semi-structured interviews completed at baseline and 8-week follow-up | Baseline and 8-week follow-up
  At the very beginning of Visit 1 and at the end of Visit 2, a random sub-sample of 15 participants from the movr group participated in semi-structured interviews that were recorded using an audio recording device (Sony ICD PX333 Digital Voice Recorder). Interview questions addressed general beliefs about fitness mobile apps and perceptions of fitness and physical functioning, individual experiences with using the movr app, how exercise perceptions may change from before to after using the movr app, and how to optimize future design and delivery of the movr app

OTHER OUTCOMES:
Changes from baseline in moderate-to-vigorous physical activity at 8-week follow-up | Baseline and 8-week follow-up
  Participants' physical activity levels were measured using the International Physical Activity Questionnaire - Short Form (IPAQ-SF)
Anthropometric measures completed at baseline and 8-week follow-up | Baseline and 8-week follow-up
  Participants' height and body mass was assessed using a stadiometer
Changes from baseline in movr Movement Assessment scores at 4- and 8-week follow-up | Baseline, and 4- and 8-week follow-up
  Participants were instructed to complete the 10 self-reported Movement Assessment tests through their individual movr app account. These movement tests are performed to assess mobility, motor control, and strength, and are used to determine deficiencies in movement patterns and to provide prescriptive information for exercise selection within the app. Participants were prompted (via email) to complete their Movement Assessments again at 4 and 8 weeks
movr app usage data measured across 8-week study period and over 8-12-week voluntary follow-up | Across 8 week study period and over 8-12 week voluntary app usage period
  The number of Minis and Builder sessions completed per week were recorded on the movr database server over the 8 week study period and additional voluntary use from 8-12 weeks
movr app usability and acceptability measured at 8-week follow-up | 8-week follow-up
  At the Visit 2 follow-up testing, participants were asked to respond to a series of Likert-type scale questions corresponding to the usability and acceptability of the movr app over the 8-week intervention period. In addition, questions included in the semi-structured interviews were also used to evaluate the usability and acceptability of the movr app

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Jung, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Diabetes Prevention Research Group Laboratory, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stork MJ, Bell EG, Jung ME. Examining the Impact of a Mobile Health App on Functional Movement and Physical Fitness: Pilot Pragmatic Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 May 28;9(5):e24076. doi: 10.2196/24076. PMID 34047704